CLINICAL TRIAL: NCT04417556
Title: Validation of Sleep Assessment Tools in the Surgical Intensive Care Unit: Comparison of Thai Version of Richards-Campbell Sleep Questionnaire, Actigraphy, and Polysomnography
Brief Title: Validation of Various Sleep Assessment Tools in SICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Annop Piriyapatsom, MD, Associate Professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 103/2563(IRB2)
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Sleep; Sleep Disturbance; Sleep Deprivation; Polysomnography; Surveys and Questionnaires; Intensive Care Unit; Adult
Keywords: Sleep Disturbance; Sleep Measurement Tools; Polysomnography; Actigraphy; Richards Campbell Questionnaire; Validation; Surgical Intensive Care Unit
MeSH Terms: conditions — Parasomnias; Sleep Deprivation | interventions — Polysomnography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep Measurement (Experimental): Sleep Measurement arm, sleep are simultaneously measured using polosomgraphy, actigraphy and Thai-version Richards Campbell Sleep Questionnaire.
  Interventions: Diagnostic Test: Sleep measurement

INTERVENTIONS:
Diagnostic Test: Sleep measurement — Sleep measurement with polysomnography, actigraphy, and Thai-version Richards Campbell Sleep Questionnaire.

SUMMARY:
Sleep deprivation is common in critical patients and it can cause impair consolidation of memory, cognitive function, metabolic function, immune, neurological and respiratory system as well as worsen the quality of life after discharge. It has been demonstrated that reducing sleep disturbance could attenuate the development of delirium in ICU patients. However, sleep evaluation is only personal perception. There are various methods for sleep monitoring, in which the most commonly mentioned methods include polysomnography, actigraphy, and the Richards-Campbell Sleep Questionnaire (RCSQ). The aims of this study is to validate the accuracy of the Thai-version RCSQ and actigraphy for sleep measurement compared to polysomnography, which is considered as the gold-standard in Thai critically ill patients admitted to surgical intensive care unit.

DETAILED DESCRIPTION:
Sleep is a periodic, reversible state of reduced consciousness, and response to external stimuli. A total sleep duration of normal human sleep is approximately 7-8 hours per night. Sleep deprivation is common in critical patients and it can cause impair consolidation of memory, cognitive function, metabolic function, immune, neurological and respiratory system as well as worsen the quality of life after discharge. The impact of sleep deprivation in critically ill patients is gaining attention as it links between sleep loss and delirium. It has been demonstrated that reducing sleep disturbance could attenuate the development of delirium in ICU patients. However, sleep evaluation is only personal perception and the previous study expressed that medical personnel evaluation still showed some error in approximately 56%. There are various methods for sleep monitoring, in which the most commonly mentioned methods include polysomnography, actigraphy, and the Richards-Campbell Sleep Questionnaire (RCSQ). Polysomnography is considered as the gold standard for monitoring the quantity and quality of sleep. Although, it is difficult to apply in critical care as it requires expensive setup and maintenance and is prone to patient dislodgment and electrical interference leading to low quality of signals and missed interpretation.

Nowadays, actigraphy has been used to assess patterns of rest and activity, which can distinguish sleep from wakefulness. The advantage of actigraphy is easy to use and non-invasive, can be used by non-specialists, and allows continuous measurement over days to weeks. On the other hand, its disadvantages are such as neuromuscular weakness and increases risk of overestimating sleep quantity as periods of inactivity scored as sleep. However, the technology has been improved recently leading to more accurate sleep measurement. Although it has been shown that actigraphy is a good alternative sleep measure in non-ICU patients, the accuracy of actigraphy is unknown in ICU patients.

For subjective tool for evaluating sleep, the Richards-Campbell Sleep Questionnaire (RCSQ) is one of the most commonly used questionnaires. It contains a simple five-item questionnaire which are sleep depth, ability to fall asleep, number of awakening, ability to fall asleep when awake and quality of sleep. The RCSQ shows a good correlation with polysomnography in sleep efficacy index. The advantages of RCSQ are easy-to-use, inexpensive and providing good quality of sleep assessment. It has been widely used in the United States and many countries. Moreover, it has been translated to many languages, such as Spanish, Swedish, German, and Japanese; and the translated version of RCSQ can be used as an alternative sleep measurement to polysomnography. Currently, our research group is translating the RCSQ into Thai version by using standard guidelines on the translation process. In spite of this, The Thai version of RCSQ (T-RCSQ) has not been validated with polysomnography before.

The aims of our study are to validate the accuracy of the T-RCSQ for sleep measurement compared to polysomnography, which is considered as the gold-standard and to access the accuracy of actigraphy for monitoring sleep quality and quantity compared to polysomnography in Thai critically ill patients admitted to surgical intensive care unit (SICU).

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years old.
* Patients who are anticipated to stay in surgical intensive care unit at least one full night (from 8 p.m. to 6 a.m. next day).
* Patients who can answer the questionnaires and can communicate, read and write in Thai.

Exclusion Criteria:

* Patients with severe cognitive impairment, dementia, Richmond Agitation Sedation Scale (RASS) score of less than -2 or more than +1 or those receiving neuromuscular blocking agents.
* Patients with pathological lesions that preclude applying electrodes and sensors of polysomnography or applying actigraphy.
* Patients with high acuity of illness whose ICU survival is not expected.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Total sleep time measured using polosomnography | 10 hours
  Total sleep time measured using polysomnography from 8 pm until 6 am next day
Total sleep time measured using wrist actigraphy | 10 hours
  Total sleep time measured using wrist actigraphy from 8 pm unitl 6 am next day
Sleep measurement using Thai-version Richards Campbell Sleep Questionnaire | 10 hours
  Sleep measurement using five-item, visual analogue scale, Thai-version Richards Campbell Sleep Questionnaire, which range from 0 to 100 mm and the higher scores indicate a better quality of sleep.

SECONDARY OUTCOMES:
Number of patients with sleep deprivation | 10 hours
  Number of patients with sleep deprivation, which is defined as total sleep time of less than 5 hours measured using polysomnography
Sleep efficiency measured using polysomnography | 10 hours
  Sleep efficiency measured using polysomnography from 8 pm until 6 am next day and defined as the ratio of total sleep time to time in bed.

CONTACTS AND LOCATIONS:
Overall Officials: Annop Piriyapatsom, MD, Principal Investigator — Mahidol University
Locations (1):
- Department of Anesthesiology, Faculty of medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No
There is no plan of sharing.

REFERENCES:
- [Background] Collop NA, Salas RE, Delayo M, Gamaldo C. Normal sleep and circadian processes. Crit Care Clin. 2008 Jul;24(3):449-60, v. doi: 10.1016/j.ccc.2008.02.002. PMID 18538194
- [Background] Gabor JY, Cooper AB, Crombach SA, Lee B, Kadikar N, Bettger HE, Hanly PJ. Contribution of the intensive care unit environment to sleep disruption in mechanically ventilated patients and healthy subjects. Am J Respir Crit Care Med. 2003 Mar 1;167(5):708-15. doi: 10.1164/rccm.2201090. PMID 12598213
- [Background] Mistraletti G, Carloni E, Cigada M, Zambrelli E, Taverna M, Sabbatini G, Umbrello M, Elia G, Destrebecq AL, Iapichino G. Sleep and delirium in the intensive care unit. Minerva Anestesiol. 2008 Jun;74(6):329-33. PMID 18500209
- [Background] Kamdar BB, Kamdar BB, Needham DM. Bundling sleep promotion with delirium prevention: ready for prime time? Anaesthesia. 2014 Jun;69(6):527-31. doi: 10.1111/anae.12686. No abstract available. PMID 24813131
- [Background] Weinhouse GL, Schwab RJ, Watson PL, Patil N, Vaccaro B, Pandharipande P, Ely EW. Bench-to-bedside review: delirium in ICU patients - importance of sleep deprivation. Crit Care. 2009;13(6):234. doi: 10.1186/cc8131. Epub 2009 Dec 7. PMID 20053301
- [Background] Nicolas A, Aizpitarte E, Iruarrizaga A, Vazquez M, Margall A, Asiain C. Perception of night-time sleep by surgical patients in an intensive care unit. Nurs Crit Care. 2008 Jan-Feb;13(1):25-33. doi: 10.1111/j.1478-5153.2007.00255.x. PMID 18226052
- [Background] Bourne RS, Minelli C, Mills GH, Kandler R. Clinical review: Sleep measurement in critical care patients: research and clinical implications. Crit Care. 2007;11(4):226. doi: 10.1186/cc5966. PMID 17764582
- [Background] Elliott R, McKinley S, Cistulli P, Fien M. Characterisation of sleep in intensive care using 24-hour polysomnography: an observational study. Crit Care. 2013 Mar 18;17(2):R46. doi: 10.1186/cc12565. PMID 23506782
- [Background] Knauert MP, Yaggi HK, Redeker NS, Murphy TE, Araujo KL, Pisani MA. Feasibility study of unattended polysomnography in medical intensive care unit patients. Heart Lung. 2014 Sep-Oct;43(5):445-52. doi: 10.1016/j.hrtlng.2014.06.049. Epub 2014 Jul 12. PMID 25023504
- [Background] de Souza L, Benedito-Silva AA, Pires ML, Poyares D, Tufik S, Calil HM. Further validation of actigraphy for sleep studies. Sleep. 2003 Feb 1;26(1):81-5. doi: 10.1093/sleep/26.1.81. PMID 12627737
- [Background] Wolters AE, Slooter AJ, van der Kooi AW, van Dijk D. Cognitive impairment after intensive care unit admission: a systematic review. Intensive Care Med. 2013 Mar;39(3):376-86. doi: 10.1007/s00134-012-2784-9. Epub 2013 Jan 18. PMID 23328935
- [Background] Richards KC, O'Sullivan PS, Phillips RL. Measurement of sleep in critically ill patients. J Nurs Meas. 2000 Fall-Winter;8(2):131-44. PMID 11227580
- [Background] Frisk U, Nordstrom G. Patients' sleep in an intensive care unit--patients' and nurses' perception. Intensive Crit Care Nurs. 2003 Dec;19(6):342-9. doi: 10.1016/s0964-3397(03)00076-4. PMID 14637294
- [Background] Krotsetis S, Richards KC, Behncke A, Kopke S. The reliability of the German version of the Richards Campbell Sleep Questionnaire. Nurs Crit Care. 2017 Jul;22(4):247-252. doi: 10.1111/nicc.12275. Epub 2017 Feb 6. PMID 28168810
- [Background] Murata H, Oono Y, Sanui M, Saito K, Yamaguchi Y, Takinami M, Richards KC, Henker R. The Japanese version of the Richards-Campbell Sleep Questionnaire: Reliability and validity assessment. Nurs Open. 2019 Mar 28;6(3):808-814. doi: 10.1002/nop2.252. eCollection 2019 Jul. PMID 31367403
- [Background] Berry RB, Brooks R, Gamaldo C, Harding SM, Lloyd RM, Quan SF, Troester MT, Vaughn BV. AASM Scoring Manual Updates for 2017 (Version 2.4). J Clin Sleep Med. 2017 May 15;13(5):665-666. doi: 10.5664/jcsm.6576. No abstract available. PMID 28416048
- [Background] Bonnet MH, Arand DL. Clinical effects of sleep fragmentation versus sleep deprivation. Sleep Med Rev. 2003 Aug;7(4):297-310. doi: 10.1053/smrv.2001.0245. PMID 14505597
- [Result] Tryon WW. Issues of validity in actigraphic sleep assessment. Sleep. 2004 Feb 1;27(1):158-65. doi: 10.1093/sleep/27.1.158. PMID 14998254